CLINICAL TRIAL: NCT01707732
Title: Adjusted Value of Thromboprophylaxis in Hospitalized Obese Patients: A Comparative Study of Two Regimens of Enoxaparin
Acronym: ITOHENOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/056/HP; 2012-001414-42 (EudraCT Number)
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Thromboprophylaxis in Hospitalized Obese Patients
Keywords: Obesity; thromboprophylaxis; Enoxaparin
MeSH Terms: conditions — Obesity | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enoxaparin 40mg/ day (Active Comparator): Enoxaparin administrated at the following dose : 40mg/ day
  Interventions: Drug: Enoxaparin
- Enoxaparin 60 mg/day (Experimental): Enoxaparin administrated at the following dose : 60 mg/day
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Administration of Enoxaparin

SUMMARY:
Venous thromboembolism (VTE), deep vein thrombosis (DVT) or pulmonary embolism (PE) is a common medical condition encountered during hospitalization in a medical environment. The use of thromboprophylaxis with Low Molecular Weight Heparin (LMWH) or fondaparinux has reduced more than 50% relative risk of thromboembolic complications.However, while obesity defined by a body mass index (BMI) greater than 30 kg/m2, is a major risk factor for venous thrombotic events, data on obese patients are limited. In fact, less than 20% of patients included in the three major studies of preventive medicine had a BMI ≥ 30 kg/m2 and most studies specific to the obese population comes from a series of bariatric surgery patients or orthopedic surgery. The main results of this series show regarding the obese population a decrease of the anti-Xa activity during the administration of a standard dose of enoxaparin (40 mg / d). However, no specific recommendation in this population has not been published to date and therefore,the dosages currently used are the same regardless of the patient's weight. In this context, the use in obese patients hospitalized in a medical environment a stronger dosage of enoxaparin (60 mg / d) compared to the standard dose of 40 mg / day, could get rates anti-Xa activity levels more consistent with the treatment required, and thus reduce the risk for thromboembolic complications in these patients

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged ≥ 18 ans.
2. Signed inform consent
3. Obesity defined by a BMI value ≥ 30 kg/m2.
4. Hospitalized for :

   * acute medical affection such as :

     * congestive heart failure (stage III or IV NYHA),
     * severe respiratory disease,
     * Infectious disease or acute rheumatologic disorder or inflammatory bowel disease with one or more additional risk factors, including active cancer, previous VTE, age > 75 y-o, estrogen therapy, chronic heart failure or chronic respiratory disease
   * or recent myocardial infarction(< 6 weeks), recent stroke with hemiparesis (< 15 days), previous VTE, myeloproliferative syndrome associated with one or more additional risk previously cited.
5. Affiliation to a welfare system.

Exclusion Criteria:

1. Subjects unwilling or unable to comply with study procedures
2. History of hypersensitivity to enoxaparin heparin induced thrombocytopenia
3. Previous history of heparin induced thrombopenia
4. acquired or inherited bleeding diathesis or coagulopathy,
5. Platelet count < 50.000 G/L,
6. History of clinically significant bleeding
7. Severe renal insufficiency with CrCl <30 ml/min (Cockcroft method),
8. Pregnancy or breastfeeding
9. Women without contraceptive methods
10. Severe peripheral arterial disease (Ankle blood pressure <50mm Hg)
11. Concomitant anticoagulant therapy
12. Severe psychiatric disease
13. History of disease or psychological or sensory anomaly susceptible to prevent the subject to understand indeed the conditions required for his participation to the protocol or preventing him from giving its enlightened consent
14. Person deprived of liberty by an administrative or judicial decision, or person under legal guardianship person
15. Patient participating to a trial or having participated in another medicinal trial within 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the anti- Xa activity between a standard treatment by Enoxaparin (40mg/ day) and an adapted dose of enoxaparin (60 mg/day) for thromboprophylaxis in obese patients hospitalized | 3 hours after third Eoxaparin injection

SECONDARY OUTCOMES:
Compare the occurrence of symptomatic venous thrombosis (deep venous thrombosis or pulmonary embolism) and the relevant bleeding events according to the enoxaparin treatments | All along the study (max 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Ygal BENHAMOU, MD, PHD, Principal Investigator — University Hospital, Rouen
Locations (1):
- UH Rouen, Rouen, France

REFERENCES:
- [Derived] Miranda S, Le Cam-Duchez V, Benichou J, Donnadieu N, Barbay V, Le Besnerais M, Delmas FX, Cuvelier A, Levesque H, Benhamou Y, Armengol G. Adjusted value of thromboprophylaxis in hospitalized obese patients: A comparative study of two regimens of enoxaparin: The ITOHENOX study. Thromb Res. 2017 Jul;155:1-5. doi: 10.1016/j.thromres.2017.04.011. Epub 2017 Apr 12. PMID 28460259